CLINICAL TRIAL: NCT01736787
Title: Efficacy and Safety of Cauliflower Mushroom Extract on Promotion of Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HANABIO-PI-CM
Record Dates: First submitted 2012-11-20; First posted 2012-11-29 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Immunity
Keywords: Cauliflower Mushroom extract; immunity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cauliflower Mushroom extract (Experimental)
  Interventions: Dietary Supplement: Cauliflower Mushroom extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cauliflower Mushroom extract — Cauliflower Mushroom extract (1g/day)
  Arms: Cauliflower Mushroom extract
Dietary Supplement: Placebo — Placebo (1g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Cauliflower Mushroom extract on promotion of immunity. The investigators measured promotion of immunity parameters , including Cytotoxicity, Cytokine (IL-4, IL-10, IFN- γ, TNF-α), and CBC (WBC, RBC, Hb, Hct, MCV, MCH, MCHC, PLT), and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 30-65 years old
* Weight within ±30% of ideal body weight
* Able to give informed consent

Exclusion Criteria:

* WBC concentration below 3000 ㎕
* Allergic or hypersensitive to any of the ingredients in the test products
* Diagnosed of gastrointestinal disease such as Immune-related diseases, severe hepatic, renal failure, and diabetes
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2013-01-18 (Actual); Study Completion 2013-01-18 (Actual)

PRIMARY OUTCOMES:
Changes in Cytotoxicity | 12 weeks
  Cytotoxicity was measured in study visit 1(0 week) and visit 3(12 week). cytotoxicity was measured by NK cell activity. Cytotoxicity (%) = (experimental release - spontaneous release) / (maximum release - spontaneous release) x 100
Changes in Cytokine (IL-4, IL-10, IFN- γ, TNF-α) | 12 weeks
  Cytokine (IL-4, IL-10, IFN- γ, TNF-α) was measured in study visit 1(0 week) and visit 3(12 week).

SECONDARY OUTCOMES:
Changes in CBC (WBC, RBC, Hb, Hct, MCV, MCH, MCHC, PLT) | 12 weeks
  CBC (WBC, RBC, Hb, Hct, MCV, MCH, MCHC, PLT) was measured in study visit 1(0 week) and visit 3(12 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea